CLINICAL TRIAL: NCT01713075
Title: Symbicort Turbuhaler 30/60 Special Clinical Experience Investigation for Long-term Use for COPD Patients
Brief Title: Symbicort Turbuhaler 30/60 Special Clinical Experience Investigation for Long-term Use for Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D589DL00001
Record Dates: First submitted 2012-10-19; First posted 2012-10-24 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; Symbicort; long-term use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Symbicort

SUMMARY:
The purpose of the investigation is to confirm the safety and efficacy in long-term use of Symbicort Turbuhaler in patients with Chronic obstructive pulmonary disease (COPD) under the post-marketing actual use.

DETAILED DESCRIPTION:
Symbicort Turbuhaler 30/60 Special Clinical Experience Investigation for long-term use for COPD patients

ELIGIBILITY:
Inclusion Criteria:

* Among patients treated with Symbicort Turbuhaler due to chronic obstructive pulmonary disease(COPD), those who received the drug for the first time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Among patients treated with Symbicort Turbuhaler due to chronic obstructive pulmonary disease(COPD), those who received the drug for the first time
Sampling Method: Non-Probability Sample
Enrollment: 1183 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | 1 year

SECONDARY OUTCOMES:
Clinical questionnaire about chronic obstructive pulmonary disease(CCQ) | At baseline, Week 12, Week 26, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — Astrazeneca KK
Locations (47):
- Japan (47):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=546&filename=D589DL00001_CSR.pdf